CLINICAL TRIAL: NCT05575661
Title: Correlation Between Postprandial Hypotension and Perioperative Adverse Events Such as Post-induction Hypotension in the Elderly: a Prospective Observational Study.
Brief Title: Correlation Between Postprandial Hypotension and Post-induction Hypotension in the Elderly.
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: I-22PJ008
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Postprandial Hypotension; Post-induction Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postprandial hypotension group: Patients who have a fall in systolic blood pressure of >20 mm Hg, or a decrease to ≤90 mm Hg when preprandial systolic blood pressure is ≥100 mm Hg within 2 hours of the lunch
- No postprandial hypotension group: Patients who do not meet the postprandial hypotension criteria within 2 hours of the lunch

SUMMARY:
Postprandial hypotension (PPH) and post-induction hypotension (PIH) are very common in the elderly population and are associated with a variety of poor outcomes.The purpose of this study is to investigate the correlation between PPH and perioperative adverse events such as PIH in the elderly.

DETAILED DESCRIPTION:
With the deepening of the aging population in our country, the number of elderly patients undergoing surgery is also increasing. Elderly patients are at higher risk for hemodynamic instability due to organ dysfunction, decreased physiological reserve, and the coexistence of multiple chronic diseases.Postprandial hypotension (PPH) is common but often unrecognized among the elderly.PPH is defined as a fall in systolic blood pressure of >20 mm Hg, or a decrease to ≤90 mm Hg when preprandial systolic blood pressure is ≥100 mm Hg within 2 hours of a meal.The pathophysiology of PPH is not clear, the decreased cardiovascular autonomic function may play an important role. Post-induction hypotension (PIH) occurs after induction but before surgical incision and autonomic dysfunction is regarded as one of the major mechanisms.This study aims to prospectively explore the correlation between PPH and perioperative adverse events such as PIH in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (≥ 65 years old）;
2. Patients with American Society of Anesthesiologists(ASA) grade I-III;
3. Patients scheduled to undergo elective non-cardiac surgery under general anesthesia, with an anticipated surgical duration of over 1 hour；
4. Patients with intra-tracheal intubation following intravenous general ；anesthesia induction and maintenance；

Exclusion Criteria:

1. Patients with vascular diseases such as aortic aneurysm, aortic dissection, symptomatic atherosclerotic obliterans, Buerger's disease, and Raynaud's syndrome
2. Patients with secondary hypertension, including renal hypertension and endocrine hypertension.
3. Patients with chronic kidney disease requiring dietary restrictions or dialysis.
4. Patients with Parkinson's disease or other conditions causing tremors.
5. Patients with problems related to oral food ingestion or those requiring enteral nutrition.
6. Patients with difficulties in measuring the upper extremities or communication problems that would interfere with study procedures.
7. Patients unable to remain in a supine position for at least 2 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients scheduled for elective non-cardiac surgery under general anesthesia in Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-induction hypotension | Within 20 minutes after induction or before incision.
  which is defined as systolic blood pressure (SBP) <90 mm Hg or a decrease of more than 30% from baseline blood pressure, mean arterial pressure(MAP)<65 mm Hg or a decrease of more than 30% from baseline blood pressure within 20 minutes after induction or before incision.

SECONDARY OUTCOMES:
Postoperative complications | Within 30 days after surgery
  We will use the Clavien-Dindo system to grade postoperative complications.
early intraoperative hypotension （eIOH） | within the first 30 minutes after the start of surgery
  which is defined asa systolic blood pressure <90 mmHg, mean arterial pressure <65 mmHg, or a decrease of more than 30% from baseline
mortality within 30 days after surgery | within 30 days after surgery
  we will assess the mortality by postoperative follow-up
12-item World Health Organization Disability Assessment Schedule 2.0 score (12-item WHODAS 2.0 score) | within 180 days after surgery
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) will be employed to evaluate postoperative functional health status. The 12-item version yields a total score ranging from 12 to 60, with higher scores indicating greater disability and poorer health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li T, Zang H, Che L, Cui Q, Xu L. Correlation between postprandial hypotension and post-induction hypotension in the elderly: a protocol for a prospective cohort study. BMJ Open. 2025 May 30;15(5):e095466. doi: 10.1136/bmjopen-2024-095466. PMID 40447437